CLINICAL TRIAL: NCT01857908
Title: A Correlative Study of Biomarkers of Resistance in Patients With Castrate Resistant Prostate Cancer Treated With Abiraterone
Status: Completed | Type: Observational
Sponsor: University Health Network, Toronto (Other)
Responsible Party: Sponsor
Other Study IDs: ABI Correlative Study; 12-5042-CE (Other: Janssen Inc.)
Record Dates: First submitted 2013-03-19; First posted 2013-05-20 (Estimated); Last update posted 2015-06-22 (Estimated); Status verified 2015-06

CONDITIONS: Prostate Cancer (Adenocarcinoma)
Keywords: Adenocarcinoma; Abiraterone; Abiraterone Acetate; Zytiga; Correlative study; Castrate Resistant Prostate Cancer; Abiraterone Correlative study
MeSH Terms: conditions — Prostatic Neoplasms; Adenocarcinoma

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective

GROUPS / COHORTS (1):
- Abiraterone acetate: All patients will be receiving abiraterone acetate as per standard of care

SUMMARY:
Adrenal androgens are serum biomarkers of interest that may help guide abiraterone acetate treatment, particularly at the time of progression. Biomarkers may also help identify pathways to resistance of abiraterone acetate treatment. The most practical way of approaching this question is to explore surrogate biomarkers of prostate cancer including quantification of pharmacodynamic endocrine biomarkers.

DETAILED DESCRIPTION:
Goals of this study include:

* Explore which circulating endocrine markers or endocrine related markers have the best potential to predict clinical response to abiraterone acetate in CRPC patients
* Explore the utility of microRNA, circulating DNA and exosome analyses in complementing the previous objective

ELIGIBILITY:
Inclusion Criteria:

* Signed written informed consent. Before any study procedures are performed, subjects (or their legally acceptable representatives) will have the details of the study described to them, and they will be given a written informed consent document to read. If subjects consent to participate in the study, they will indicate that consent by signing and dating the informed consent document in the presence of study personnel
* Be suitable for receiving treatment with abiraterone acetate and prednisone
* Patients must have histologically or cytologically confirmed adenocarcinoma of the prostate without neuroendocrine differentiation or small cell histology
* Patients may not receive any other investigational agent or dose escalation of abiraterone acetate during study participation
* Patient consents to comply to treatment with abiraterone acetate as directed by their physician

Exclusion Criteria:

* Taking a dose of abiraterone acetate other than 1g daily or lack of compliance to daily dosing of abiraterone acetate and prednisone
* Patients receiving spironolactone or any other steroidogenic compounds in excess of the associated prednisone 5mg bid are excluded due to the potential for androgen receptor agonism

Sex: Male | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients receiving Abiraterone Acetate for Castrate Resistant Prostate Cancer
Sampling Method: Non-Probability Sample
Enrollment: 20 (Actual)
Dates: Start 2012-06; Primary Completion 2014-11 (Actual)

PRIMARY OUTCOMES:
PSA | Patients will be followed from Day 1 (date of initiation of Abiraterone treatment) until the date of first documented progression (estimated to be 1 year). PSA will be assessed every 30 days (approximately) until the time of PSA/clinical progression
  PSA nadir samples will be assessed and compared to pre-Abiraterone treatment samples post completion of study

CONTACTS AND LOCATIONS:
Overall Officials: Anthony Joshua, BSc(Med) MBBS PhD FRACP, Principal Investigator — Princess Margaret Cancer Centre; Bernie Eigl, MD, Principal Investigator — British Columbia Cancer Agency
Locations (2):
- Canada (2):
  - BC Cancer Agency, Vancouver, British Columbia
  - Princess Margaret Cancer Centre, Toronto, Ontario